CLINICAL TRIAL: NCT02296983
Title: A Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of the BPSC1001 (VSVΔG-ZEBOV) Ebola Virus Vaccine Candidate in Healthy Adult Volunteers in Kilifi, Kenya.
Brief Title: A Study to Find Out if the New Ebola Vaccine is Safe and Stimulates Immunity That Might Protect Adults in Kilifi, Kenya.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: World Health Organization (Other); Wellcome Trust (Other); Institute of Tropical Medicine, University of Tuebingen (Other); Albert Schweitzer Hospital (Other); Philipps University Marburg (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OXTREC 71-14; SSC 2976 (Other: KEMRI Scientific Steering Committee)
Record Dates: First submitted 2014-11-11; First posted 2014-11-21 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose arm (Experimental): The low dose cohort will receive an intramuscular (deltoid) injection of 3x106 pfu of VSV-ZEBOV vaccine.
  Interventions: Biological: VSV-ZEBOV
- Full dose arm (Experimental): The full dose cohort will receive an intramuscular (deltoid) injection1x107 pfu of VSV-ZEBOV vaccine.
  Interventions: Biological: VSV-ZEBOV

INTERVENTIONS:
Biological: VSV-ZEBOV — VSV-ZEBOV
  Other Names: BSPSC1001

SUMMARY:
Previous Ebola outbreaks have been limited to individual countries and contained by infection control activities. The current outbreak in West Africa is international, and air travel has resulted in a number of infected travellers crossing national borders. There are currently no specific treatments generally available for Ebola and the mortality is high, particularly in countries with limited intensive care facilities. There is currently no vaccine and the personal protection required by healthcare workers treating patients is cumbersome and requires full compliance to be protective.

There is now a consortium (VEBCON collaboration) of four clinical centres (in Kenya, Gabon, Switzerland and Germany), WHO and New Link Genetics (the vaccine manufacturer) under which this study will be conducted. The investigators are conducting this trial, a Phase I, open-label, dose escalation trial, designed to establish safety, tolerability and immunogenicity of two doses of VSVΔG-ZEBOV, an Ebola Virus Vaccine Candidate for the first time in sub-Saharan African populations.

The investigators plan to vaccinate 40 volunteers in Kenya. The trial will be conducted at the KEMRI-CGMR Coast site where healthcare workers (both clinical and laboratory) will be the primary target population as they are likely to be the recipients of a protective vaccine. The investigators will vaccinate a cohort of 20 volunteers at a low dose and then vaccinate a further cohort of 20 volunteers at full dose. Each volunteer will receive one dose of the vaccine. The investigators will follow them up for a period of one year looking to their safety and immunogenicity endpoints.

DETAILED DESCRIPTION:
This study is being conducted to assess safety and immunogenicity of an experimental ebola vaccine.

An outbreak due to the Ebola Zaire (ZEBOV) strain of unprecedented magnitude and scope and with a high mortality continues to spread across West Africa. No vaccine is currently licensed.

The specific opportunity at hand with rVSVΔG-ZEBOV-GP (BPSC1001) is to achieve long-lasting protective immunity to ZEBOV on a time scale of weeks in humans upon a single-shot vaccination, offering a discrete benefit over prime-boost vaccination protocols. The current outbreak represents a global health emergency and the need for access to therapeutic intervention and vaccines is paramount.

The vaccine investigated in this study might provide a critical tool to suppress future out-breaks of EVD in areas at risk.

This study is 1 of 4 clinical trials currently conducted as part of the WHO-led VEBCON consortium, aiming to generate harmonized data for the rVSVΔG-ZEBOV-GP (BPSC1001) vaccine candidate to allow optimized rapid decisions on dose and safety.

ELIGIBILITY:
Inclusion Criteria:

* • Have provided written informed consent prior to screening procedures (i.e. participants must be literate).

  * Healthy adult male or non-pregnant, non-lactating female, ages 18 to 55 (inclusive) at the time of screening
  * Free of clinically significant health problems, as determined by pertinent medical history, clinical examination and blood tests at screening
  * Available, able, and willing to participate for all study visits and procedures
  * Negative pregnancy-test for female volunteers
  * Females, of non-childbearing potential who are post-menopausal (i.e. ≥ one year without menses) or surgically sterilized (tubal ligation, bilateral oophorectomy, or hysterectomy)
  * Females, of childbearing potential, who are willing to use effective methods of contraception for 14 days before vaccination and 30 days after vaccination.
  * Males who are willing to use effective contraception following vaccination for a period of one week.
  * Be willing to minimize blood and body fluid exposure of others for 5 days after vaccination

Exclusion Criteria:

* • History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions.

  * Known allergy to the components of the BPSC1001 vaccine product
  * Unable or unwilling to stay in the study area for the period of the study and comply with study procedures.
  * Ongoing participation in another clinical trial
  * Receipt of licensed vaccines within 14 days of planned study immunization (30 days for live vaccines)
  * Acute or chronic, clinically significant psychiatric, hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical exam, and/or laboratory screening test
  * Any serologic evidence of hepatitis B SAg or HIV infection.
  * Any confirmed or suspected immunosuppressive or immunodeficient condition, cytotoxic therapy in the previous 5 years, and/or uncontrolled diabetes
  * Have an active malignancy or history of metastatic or hematologic malignancy
  * Suspected or known alcohol and/or illicit drug abuse within the past 5 years
  * Moderate or severe illness and/or fever >38°C within 2 weeks prior to vaccination
  * Pregnant or lactating woman or a woman who intends to become pregnant within 30 days following vaccination.
  * Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
  * Administration of chronic (defined as more than 14 days) immunosuppressant's or other immune modifying drugs within 6 months of study entry
  * Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The nature, frequency, and severity of adverse events (AEs) and/or serious adverse events (SAEs) with causal link to the study intervention | Days 0-30
  To evaluate the safety and tolerability of two different doses of VSVΔG-ZEBOV vaccine

SECONDARY OUTCOMES:
Incidence and severity of local and systemic reactogenicity signs and symptoms | Day 0-28
Incidence of unsolicited adverse events (AEs) | Days 0-28
Incidence of serious adverse events (SAEs) | Days 0-365
Distribution of values of safety laboratory measures at baseline and at follow-up visits post-vaccination | Day 0-30
  The distribution of values of safety laboratory measures will include the assessment of complete blood count (with differential white cell count), creatinine and alanine transaminase levels at baseline and day 7 and 30 following vaccine administration.
Persistence of titres of ZEBOV-specific IgG antibodies | 0-180 days
Detection, magnitude and duration of VSV-ZEBOV viraemia and shedding | Day 1, 3 and 7
  The detection and concentration (copies/ml) of rVSV (viral shedding) will determined in blood, urine, or saliva samples to evaluate VSV vaccine viraemia following vaccine administration. The duration will be determined by the last timepoint with detectable viraemia.This is a composite measure.
Titres of neutralising ZEBOV-specific IgG antibodies | Days 7, 30, 60, 90, 180 and 365
Pattern of ZEBOV specific T cell responses | Days 7, 30, 90, 180 and 365
Titers of ZEBOV-specific IgG antibodies | Days 0-28
  Important for dose selection

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bejon, MD, PhD, Principal Investigator — KEMRI-Wellcome Trust Collaborative Research Program
Locations (1):
- KEMRI Wellcome Trust Research Programme, Kilifi, Coast, Kenya

REFERENCES:
- [Derived] Huttner A, Agnandji ST, Combescure C, Fernandes JF, Bache EB, Kabwende L, Ndungu FM, Brosnahan J, Monath TP, Lemaitre B, Grillet S, Botto M, Engler O, Portmann J, Siegrist D, Bejon P, Silvera P, Kremsner P, Siegrist CA; VEBCON; VSV-EBOVAC; VSV-EBOPLUS Consortia. Determinants of antibody persistence across doses and continents after single-dose rVSV-ZEBOV vaccination for Ebola virus disease: an observational cohort study. Lancet Infect Dis. 2018 Jul;18(7):738-748. doi: 10.1016/S1473-3099(18)30165-8. Epub 2018 Apr 5. PMID 29627147
- [Derived] Coller BG, Blue J, Das R, Dubey S, Finelli L, Gupta S, Helmond F, Grant-Klein RJ, Liu K, Simon J, Troth S, VanRheenen S, Waterbury J, Wivel A, Wolf J, Heppner DG, Kemp T, Nichols R, Monath TP. Clinical development of a recombinant Ebola vaccine in the midst of an unprecedented epidemic. Vaccine. 2017 Aug 16;35(35 Pt A):4465-4469. doi: 10.1016/j.vaccine.2017.05.097. Epub 2017 Jun 21. PMID 28647166
- [Derived] Medaglini D, Harandi AM, Ottenhoff TH, Siegrist CA; VSV-Ebovac Consortium. Ebola vaccine R&D: Filling the knowledge gaps. Sci Transl Med. 2015 Dec 9;7(317):317ps24. doi: 10.1126/scitranslmed.aad3106. PMID 26659569
- [Derived] Agnandji ST, Huttner A, Zinser ME, Njuguna P, Dahlke C, Fernandes JF, Yerly S, Dayer JA, Kraehling V, Kasonta R, Adegnika AA, Altfeld M, Auderset F, Bache EB, Biedenkopf N, Borregaard S, Brosnahan JS, Burrow R, Combescure C, Desmeules J, Eickmann M, Fehling SK, Finckh A, Goncalves AR, Grobusch MP, Hooper J, Jambrecina A, Kabwende AL, Kaya G, Kimani D, Lell B, Lemaitre B, Lohse AW, Massinga-Loembe M, Matthey A, Mordmuller B, Nolting A, Ogwang C, Ramharter M, Schmidt-Chanasit J, Schmiedel S, Silvera P, Stahl FR, Staines HM, Strecker T, Stubbe HC, Tsofa B, Zaki S, Fast P, Moorthy V, Kaiser L, Krishna S, Becker S, Kieny MP, Bejon P, Kremsner PG, Addo MM, Siegrist CA. Phase 1 Trials of rVSV Ebola Vaccine in Africa and Europe. N Engl J Med. 2016 Apr 28;374(17):1647-60. doi: 10.1056/NEJMoa1502924. Epub 2015 Apr 1. PMID 25830326